CLINICAL TRIAL: NCT03232957
Title: Efficacy and Side Effects of Intrathecal Morphine in Multimodal Analgesia for Unilateral Total Knee Arthroplasty
Brief Title: Intrathecal Morphine for Unilateral Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Assistant professor, Department of Anesthesiology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si 331/2017
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Primary Osteoarthritis of Knee Nos
Keywords: Intrathecal morphine, total knee arthroplasty
MeSH Terms: interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: In the anesthetic record, 0.5% isobaric bupivacaine with study drug is recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No IT morphine (Experimental): Spinal block with 0.5% isobaric with no intrathecal morphine
  Interventions: Procedure: No IT morphine; Drug: Morphine; Drug: Bupivacaine
- 50 ug IT morphine (Experimental): Spinal block with 0.5% isobaric with 50 ug intrathecal morphine
  Interventions: Procedure: 50 ug IT morphine; Drug: Morphine; Drug: Bupivacaine
- 100 ug IT morphine (Experimental): Spinal block with 0.5% isobaric with 100 ug intrathecal morphine
  Interventions: Procedure: 100 ug IT morphine; Drug: Morphine; Drug: Bupivacaine

INTERVENTIONS:
Procedure: 50 ug IT morphine — Spinal block with bupivacaine and intrathecal morphine 50 ug
  Arms: 50 ug IT morphine
Procedure: 100 ug IT morphine — Spinal block with bupivacaine and intrathecal morphine 100 ug
  Arms: 100 ug IT morphine
Procedure: No IT morphine — Spinal block with bupivacaine and intrathecal morphine 0 ug
  Arms: No IT morphine
Drug: Morphine — intrathecal morphine
Drug: Bupivacaine — 0.5 isobaric bupivacaine

SUMMARY:
This study evaluates postoperative numerical pain score and systemic opioid requirement within 48 hours for unilateral total knee arthroplasty. Comparing among 3 groups of intrathecal morphine; 0,50, 100 ug with multimodal analgesia.

DETAILED DESCRIPTION:
Intrathecal opioid is effective postoperative analgesia for orthopedic lower extremity surgery. However there are some limitations such as nausea, vomiting, pruritus, dizziness. Nowadays multimodal analgesia is used in unilateral total knee arthroplasty include oral analgesic drugs, adductor canal block and local analgesia infiltration.

This study evaluates whether intrathecal opioid should be added in the role of multimodal analgesia in total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Aged more than 18 years old undergoing unilateral total knee arthroplasty
* American Society of Anesthesiologists physical status classification 1-3

Exclusion Criteria:

* Participants deny to enroll the study
* Allergy to local anesthetics, opioid and NSAIDs
* Hepatic disease
* Contraindication for neuraxial block or adductor canal block
* Uncontrolled cardiovascular disease
* Creatinine clearance less than 50 ml/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Numerical rating scale | Within 48 hours
  Numerical rating scale 0-10

SECONDARY OUTCOMES:
Morphine requirement | Within 48 hours
  Systemic morphine requirement
Nausea vomiting | Within 48 hours
  Incidence and severity of nausea and vomiting
Pruritus | Within 48 hours
  Incidence and severity of pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stowers MD, Lemanu DP, Coleman B, Hill AG, Munro JT. Review article: Perioperative care in enhanced recovery for total hip and knee arthroplasty. J Orthop Surg (Hong Kong). 2014 Dec;22(3):383-92. doi: 10.1177/230949901402200324. PMID 25550024
- [Background] Rathmell JP, Pino CA, Taylor R, Patrin T, Viani BA. Intrathecal morphine for postoperative analgesia: a randomized, controlled, dose-ranging study after hip and knee arthroplasty. Anesth Analg. 2003 Nov;97(5):1452-1457. doi: 10.1213/01.ANE.0000083374.44039.9E. PMID 14570664
- [Background] Ibrahim MS, Alazzawi S, Nizam I, Haddad FS. An evidence-based review of enhanced recovery interventions in knee replacement surgery. Ann R Coll Surg Engl. 2013 Sep;95(6):386-9. doi: 10.1308/003588413X13629960046435. PMID 24025284
- [Background] Hassett P, Ansari B, Gnanamoorthy P, Kinirons B, Laffey JG. Determination Of The Efficacy And Side-effect Profile Of Lower Doses Of Intrathecal Morphine In Patients Undergoing Total Knee Arthroplasty. BMC Anesthesiol. 2008 Sep 24;8:5. doi: 10.1186/1471-2253-8-5. PMID 18816386
- [Background] Nakai T, Tamaki M, Nakamura T, Nakai T, Onishi A, Hashimoto K. Controlling pain after total knee arthroplasty using a multimodal protocol with local periarticular injections. J Orthop. 2013 Mar 17;10(2):92-4. doi: 10.1016/j.jor.2013.02.001. eCollection 2013. PMID 24403757
- [Background] McCartney CJ, Nelligan K. Postoperative pain management after total knee arthroplasty in elderly patients: treatment options. Drugs Aging. 2014 Feb;31(2):83-91. doi: 10.1007/s40266-013-0148-y. PMID 24399578
- [Background] Kunopart M, Chanthong P, Thongpolswat N, Intiyanaravut T, Pethuahong C. Effects of single shot femoral nerve block combined with intrathecal morphine for postoperative analgesia: a randomized, controlled, dose-ranging study after total knee arthroplasty. J Med Assoc Thai. 2014 Feb;97(2):195-202. PMID 24765899